CLINICAL TRIAL: NCT02897622
Title: Severe and Enduring Eating Disorder Patients at Stockholms Center for Eating Disorders in Sweden
Acronym: SEED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Yvonne von Hausswolff-Juhlin, Associated professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eira
Record Dates: First submitted 2016-08-12; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Eating Disorders
Keywords: Eating disorders; severe and enduring; quality of life; case management
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Case management (Other): Case management
  Interventions: Other: Case management

INTERVENTIONS:
Other: Case management — Case management by Eira unit

SUMMARY:
Patients with severe and enduring eating disorders (SEED) are seriously ill and have a low quality of life. In 2014, a special unit based on case management (CM), for patients with SEED (the Eira unit) was started at Stockholm Centre for Eating Disorders, Sweden. Eating disorder is a serious illness that creates a great deal of suffering. Most patients who undergo specialized eating disorder treatment will be healthy, but a small percentage of the patients develop a SEED. SEED patient have gone through numerous of treatments and has been to several specialists units for years as well as they has completed many different therapies without getting fee from the eating disorder (ED). Due to the long term sick in ED the SEED patient is often alone and has difficulties to cope with everyday life situations. SEED patients are a vulnerable patient population with a great suffering and poverty to release the identity of the ED. However, no previous study is done in which patients with SEED themselves describe their own theory about why they are still ill and how specialized eating disorder care has affected them. In the ED field, there is a growing consensus that treatment of patients with SEED needs to be multi-professional, with a focus on improving the patients' social situation, minimizing medical complications, and enhancing quality of life and independence, rather than focusing one-sided on symptom reduction. Is case management a way to help the SEED patients witness a better quality of life? Besides the personal suffering of patients and their families, SEED is also associated with high costs for health care and for society in general.

DETAILED DESCRIPTION:
1. This is a qualitative study based on semi-structured interviews with 21 patients with SEED. Grounded theory was used to analyse data. The patients had suffered from eating disorders on average for 21,5 years with a BMI of 15,4 (12,2-19.5) at the time for the interview.
2. Methods for data collection are a semi-structured diagnostic interview, a qualitative interview, self-report questionnaires and data from medical records. The diagnostic interview and the self-report assessments will be done at start of treatment and at follow-ups after one, two, and three years. The qualitative interview will be conducted one year after start of treatment. Data from medical records will be collected retrospectively.

The Structured Eating Disorder Interview (SEDI) is a semi-structured diagnostic interview for ED diagnoses according to the DSM-IV. The interview consists of a maximum of 30 and normally about 20-25 questions.

The RAND-36 (also known as the SF-36) measures health-related quality of life (HRQoL). Changes in the HRQoL over time can be seen by comparing repeated assessments.

The Eating Disorder Examination Questionnaire (EDE-Q) measures central symptomatic aspects of ED by way of patient's self-ratings.

The Treatment Satisfaction Scale 2 (TSS-2) is a patient-rated assessment of treatment satisfaction in a simple 6-item scale. TSS-2 will be used at all follow-ups.

The qualitative interview is semi-structured and consists of three broad themes:

1. The patient's thoughts about her/his life situation in the year he/she has been at Eira.
2. The patient's thoughts and reflections about her/his quality of life, and whether it has been affected in the year he/she has been at Eira.
3. The patient's thoughts about her/his future. The informants will be asked to talk openly around these themes. The interviewer, who is the same person for all interviews, is a psychologist who is not part of the Eira staff.

4. The cost-effectiveness analysis consists of costs of the CM intervention, changes in quality of life, as well as societal costs such as health care usage and loss of production. The perspective of the analysis will be societal and the time horizon three years. The analysis method is going to be cost-utility analysis with health effect expressed in quality adjusted life years (QALY). The analysis will be complemented with the probability of acceptable cost-effectiveness with different willingness to pay for a QALY.

All costs of the CM intervention occur at Eira. The cost for each patient in the study can be calculated by Eira's total cost divided with each patient's share of resource utilization based on enrolled time.

QALYs will be estimated based on RAND-36 transformed to SF-6D based on a British preference score. From the measures at baseline, and after 1, 2 and 3 years, changes in QALYs can be estimated. From medical records, changes in cost of health care usage can be calculated. The participants' employment and change acquisition work rate is followed during the same period based on interviews with participants.

The treatment may also have impact on relatives' quality of life, costs and earnings. These aspects will not be considered in the analysis.

Setting

During the first 5-6 sessions at Eira, the patient's psychiatric, somatic and social condition is carefully investigated as well as her/his medical history and previous treatment experiences. Thereafter the CM intervention starts. The patients' needs and preferences guides where and how often the meetings take place and some can be done by phone or text messages. Another important part of the CM is to help the patients contact the authorities and if necessary to aid them with economic issues.

In addition to the supportive interventions is it also important to regularly monitor the somatic condition and the weight of the patients. If the patient is temporarily in need of more somatic or psychiatric help, the therapists can help in planning a short, more intensive treatment.

Twice a year, there is a lecture about the SEED condition for the relatives (without the patients) at Eira. During the lecture the relatives can ask questions and discuss problems they encounter as SEED relatives. With the patients' consent, relatives are invited to participate in the CM treatment. Information and support is offered relatives on an individual basis, this also includes underage children.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis: eating disorder according to DSM IV (Diagnostic and statistical manual of mental disorders fourth edition) Criteria based on diagnostic interview
* Illness duration of ED >10
* Participated in at least three failed specialized eating disorder treatments
* Written informed consent
* Having the mental capacity to make provide informed consent to research participation
* Somatically stable

Exclusion Criteria:

* Somatically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-04; Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Patients experience of specialized eating disorder care | up to 5 years
  By semi structured interviews

SECONDARY OUTCOMES:
Quality of life | up to 5 years
  RAND-36
Cost-effectiveness | up to 5 years
  RAND-36

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne von Hausswolff-Juhlin, MdPhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Maja Molin, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Molin M, von Hausswolff-Juhlin Y, Norring C, Hagberg L, Gustafsson SA. Case management at an outpatient unit for severe and enduring eating disorder patients at Stockholm Centre for Eating Disorders- a study protocol. J Eat Disord. 2016 Oct 26;4:24. doi: 10.1186/s40337-016-0121-3. eCollection 2016. PMID 27800159